CLINICAL TRIAL: NCT04530188
Title: Effects of Sevoflurane on Extravascular Lung Water and Pulmonary Vascular Permeability in Patients With Acute Respiratory Distress Syndrome
Brief Title: Effects of Sevoflurane on Extravascular Lung Water and Pulmonary Vascular Permeability in Patients With ARDS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Christopher Lai, principal investigator, Bicetre Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BicetreH
Record Dates: First submitted 2020-08-14; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: ARDS; ARDS, Human
Keywords: ARDS; inhaled anesthetic; sevoflurane; extravascular lung water; pulmonary vascular permeability
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhaled sedation with sevoflurane (Experimental): Inhaled sedation with sevoflurane using the Anesthesia Conserving Device (AnaConDa-S, Sedana Medical, Danderyd, Sweden)
  Interventions: Drug: Sevoflurane
- intravenous sedation with propofol (Active Comparator): intravenous sedation with propofol, as already used in our ICU
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Inhaled sedation with sevoflurane using the Anesthesia Conserving Device (AnaConDa-S, Sedana Medical, Danderyd, Sweden)
  Arms: inhaled sedation with sevoflurane
Drug: Propofol — Intravenous sedation with propofol, as already used in our ICU
  Arms: intravenous sedation with propofol

SUMMARY:
The study will investigate the effects of inhaled sedation with sevoflurane using the AnaConDa device on extravascular lung water index (EVLWi) and the pulmonary vascular permeability index (PVPI) in patients with moderate to severe acute respiratory distress syndrome (ARDS). Improvement in oxygenation and decreases in lung inflammatory response has been demonstrated in patients with ARDS compared with intravenous sedation. However, preclinical data showing a decrease in lung edema has not been confirmed. The hypothesis is that inhaled sedation with sevoflurane reduces EVLWi and PVPI in patients with ARDS, assessed with the PiCCO device. Patients will receive either inhaled sedation (interventional group), or a sedation with propofol (control group). Both will be associated with remifentanil. Sedation will be monitored by bispectral index with a targeted value of 30-50. The primary outcome will be daily assessment of EVLWi and PVPI over time in patients sedated with sevoflurane compared to propofol. Secondary outcomes will include value of PVPI and EVLW at 48h after intubation, fluid administration, need in norepinephrine, time between cessation of sedation and trial of weaning sedation, ventilation free days, mortality at day 28, the partial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2), plasma and alveolar levels of cytokines (tumor necrosis factor (TNF)-α, interleukine (IL)-1β, IL-6, IL-8). These blood and alveolar samples will be done at baseline, on day 2 and on day 5. A sub-group analysis will be done in Covid-19 related ARDS. Decrease in PVPI and EVLWi with inhaled sevoflurane may be related to the decrease in lung edema in ARDS patients and may ultimately improve patient outcome.

DETAILED DESCRIPTION:
Background:

Inhaled sedation with volatile anesthetic agents has been proposed as an efficient and safe alternative to usual intravenous sedation such as propofol or midazolam in the intensive care unit. In acute respiratory distress syndrome (ARDS) models, preclinical studies comparing inhaled sedation to intravenous sedation showed that sedation with sevoflurane improves oxygenation, reduces the lung and systemic inflammatory response, decreases formation of alveolar edema and is associated with a less pronounced increase in extravascular lung water (EVLW, the amount of water contained in the lungs outside the pulmonary vasculature) or pulmonary vascular permeability index (PVPI), the ratio of EVLW over the pulmonary blood volume). Although benefits of inhaled sedation on inflammation and oxygenation have been shown in humans, its direct effect on EVLW or PVPI has never been evaluated in patients with ARDS. It could be important as their levels are factors independently associated with mortality in patients with ARDS.

Aim:

To evaluate the effect of inhaled sedation with sevoflurane in comparison with sedation with propofol on the degree of PVPI and the amount of EVLW in patients with moderate-to-severe ARDS.

Hypothesis:

The hypothesis is that inhaled sedation with sevoflurane reduces PVPI and EVLW in patients with ARDS compared to sedation with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of acute respiratory distress syndrome for ≤24 hours of all of the following conditions, within one week of a clinical insult or new or worsening respiratory symptoms:
* PaO2/FiO2 <150 mmHg with positive end-expiratory pressure (PEEP) ≥8 cmH2O (or, if arterial blood gas not available, SpO2/FiO2 that is equivalent to a
* PaO2/FiO2 <150 mmHg with PEEP ≥8 cmH2O and a confirmatory SpO2/FiO2 between 1-6 hours after the initial SpO2/FiO2 determination)
* Bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules
* Respiratory failure not fully explained by cardiac failure or fluid overload; need objective assessment (e.g., echocardiography) to exclude hydrostatic edema if no risk factor present
* PaO2/FiO2 <200 mmHg after meeting inclusion criteria and before randomization

Exclusion Criteria:

* Absence of affiliation to the French Sociale security
* Patient under a tutelage measure or placed under judicial protection
* Known pregnancy
* Currently receiving ECMO therapy
* Chronic liver disease defined as a Child-Pugh score of 12-15
* Severe hepatic failure
* Expected duration of mechanical ventilation <48 hours
* Moribund patient, i.e. not expected to survive 24 hours despite intensive care Burns >70% total body surface
* Previous hypersensitivity or anaphylactic reaction to sevoflurane
* Medical history of malignant hyperthermia
* Medical history of liver disease attributed to previous exposure to a halogenated agent
* Known hypersensitivity to propofol or any of its components
* Suspected or proven intracranial hypertension
* Tidal volume of 6 mL/kg predicted body weight (PBW) below 200 mL (as recommended by the manufacturer for the use of the AnaConDa-S (Sedana Medical, Danderyd, Sweden)
* Enrollment in another interventional ARDS trial with direct impact on sedation and mechanical ventilation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Time course of extravascular lung water (EVLW) | Through study completion, up to 90 days
  EVLW is the amount of water contained in the lungs outside the pulmonary vasculature. It can be measured using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Time course of pulmonary vascular permeability index (PVPI) | Through study completion, up to 90 days
  PVPI is estimated using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)

SECONDARY OUTCOMES:
Value of extravascular lung water index (EVLW) | Day 2
  EVLW is the amount of water contained in the lungs outside the pulmonary vasculature. It can be measured using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Value of extravascular lung water index (EVLW) | Day 5
  EVLW is the amount of water contained in the lungs outside the pulmonary vasculature. It can be measured using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Value of pulmonary vascular permeability index (PVPI) | Day 2
  PVPI is estimated using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Value of pulmonary vascular permeability index (PVPI) | Day 5
  PVPI is estimated using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Daily fluid balance | Through study completion, up to 90 days
  Fluid balance will be calculated daily as fluid intake minus fluid output. It is expressed in mL/day.
Need in catecholamines | Through study completion, up to 90 days
time between sedation cessation and first weaning trial | Through study completion, up to 90 days
Ventilator free days | Day 28
  ventilator-free days to taking into account death as a competing event
Mortality | Day 28
Oxygenation assessed with PaO2/FiO2 ratio | Day 2
Oxygenation assessed with PaO2/FiO2 ratio | Day 5
Oxygenation assessed with PaO2/FiO2 ratio | Through study completion, up to 90 days
Plasma and alveolar levels of proinflammatory cytokines : tumor necrosis factor alpha (TNFα, interleukin (IL)-1β, IL-6, IL-8 | At enrollment
  Blood samples and alveolar samples from a bronchoalveolar lavage to constitute a biological collection aimed at further investigating the effects of inhaled sedation with sevoflurane in patients with ARDS
Plasma and alveolar levels of proinflammatory cytokines : tumor necrosis factor alpha (TNFα, interleukin (IL)-1β, IL-6, IL-8 | Day 2
  Blood samples and alveolar samples from a bronchoalveolar lavage to constitute a biological collection aimed at further investigating the effects of inhaled sedation with sevoflurane on inflammation in patients with ARDS
Plasma and alveolar levels of proinflammatory cytokines : tumor necrosis factor alpha (TNFα, interleukin (IL)-1β, IL-6, IL-8 | Day 5
  Blood samples and alveolar samples from a bronchoalveolar lavage to constitute a biological collection aimed at further investigating the effects of inhaled sedation with sevoflurane on inflammation in patients with ARDS
Cardiac index | Through study completion, up to 90 days
  Data provided by transpulmonary thermodilution. (unit: L/min/m2)
Global End Diastolic Volume index | Through study completion, up to 90 days
  Data provided by transpulmonary thermodilution. (unit: mL/m2)
Blood pressure | Through study completion, up to 90 days
  Systolic, diastolic and mean blood pressure
Correlation between data provided by transpulmonary thermodilution (extravascular lung water, pulmonary vascular permeability index, cardiac index, global end-diastolic volume) and 28-day mortality | up to 28 days
  maximal or minimal values, trend in values,

IPD SHARING:
Plan to Share IPD: Undecided